CLINICAL TRIAL: NCT02767921
Title: A Pilot Study of Neoadjuvant sEphB4-HSA in Patients With Genitourinary Cancers
Brief Title: sEphB4-HSA Before Surgery in Treating Patients With Bladder Cancer, Prostate Cancer, or Kidney Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Insufficient accrual
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0S-15-6; NCI-2015-02236 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 0S-15-6 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2016-05-06; First posted 2016-05-11 (Estimated); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Infiltrating Bladder Urothelial Carcinoma; Recurrent Bladder Carcinoma; Stage I Prostate Cancer; Stage I Renal Cell Cancer; Stage II Bladder Urothelial Carcinoma; Stage II Renal Cell Cancer; Stage IIA Prostate Cancer; Stage IIB Prostate Cancer; Stage III Prostate Cancer; Stage III Renal Cell Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms; Prostatic Neoplasms; Carcinoma, Renal Cell | interventions — Cystectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (recombinant EphB4-HSA fusion protein, surgery) (Experimental): Patients receive recombinant EphB4-HSA fusion protein IV over 60 minutes once weekly for 3 weeks (3 doses) in the absence of disease progression or unacceptable toxicity. Patients who agree may receive the fourth dose after an additional week as determined by the study medical oncologist. Two to four weeks after the last dose of recombinant EphB4-HSA fusion protein, patients undergo robotic-assisted radical cystectomy or robotic-assisted radical or partial nephrectomy.
  Interventions: Other: Cytology Specimen Collection Procedure; Other: Laboratory Biomarker Analysis; Procedure: Radical Cystectomy; Biological: Recombinant EphB4-HSA Fusion Protein; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Other: Cytology Specimen Collection Procedure — Correlative studies
  Other Names: Cytologic Sampling
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Radical Cystectomy — Undergo robotic-assisted radical cystectomy
  Other Names: Complete Cystectomy
Biological: Recombinant EphB4-HSA Fusion Protein — Given IV
  Other Names: sEphB4-HSA
Procedure: Therapeutic Conventional Surgery — Undergo robotic-assisted radical or partial nephrectomy

SUMMARY:
This pilot clinical trial studies the side effects of recombinant EphB4-HSA fusion protein before surgery in treating patients with transitional cell carcinoma of the bladder, prostate cancer, or kidney cancer. Recombinant EphB4-HSA fusion protein may block an enzyme needed for tumor cells to multiply and may also prevent the growth of new blood vessels that bring nutrients to the tumor. Giving recombinant EphB4-HSA fusion protein before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility of, and adverse events associated with, treatment with soluble ephrin type-B receptor 4 (sEphB4)-human serum albumin (HSA) (recombinant EphB4-HSA fusion protein) prior to minimally invasive robotic surgery in patients with either muscle-invasive transitional cell carcinoma of the bladder; clear cell renal cell carcinoma (4 cm or greater); or prostate cancer Gleason (7 or under).

SECONDARY OBJECTIVES:

I. To determine tumor response to neoadjuvant sEphB4 as measured by imaging response and pathologic response.

TERTIARY OBJECTIVES:

I. To evaluate the expression of ephrin type-B receptor 4 (EphB4) and eph-related receptor tyrosine kinase ligand 5 (EphrinB2) in the archival tumor samples and explore potential associations with outcome.

II. To bank specimens for future correlative biomarker studies based on the results of ongoing biomarkers analyses in the phase I of sEphB4-HSA as a single agent.

III. To evaluate changes in deoxyribonucleic acid (DNA) methylation of the surgical specimen after being treated with sEphB4-HSA.

IV. To evaluate the infiltration of immune cells into the tumor due to administering sEphB4-HSA.

V. To evaluate the impact sEphB4-HSA has on vessel density on the tumor tissue. VI. To assess the applicability of using sEphB4-HSA for treating genitourinary cancers.

VII. To assess the applicability of using contrast-enhanced ultrasound imaging for determining pathological complete response (pCR) rate.

OUTLINE:

Patients receive recombinant EphB4-HSA fusion protein intravenously (IV) over 60 minutes once weekly for 3 weeks (3 doses) in the absence of disease progression or unacceptable toxicity. Patients who agree may receive the fourth dose after an additional week as determined by the study medical oncologist. Two to four weeks after the last dose of recombinant EphB4-HSA fusion protein, patients undergo robotic-assisted radical cystectomy or robotic-assisted radical or partial nephrectomy.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization for release of personal health information

  * NOTE: HIPAA authorization may be included in the informed consent or obtained separately
* Eastern Cooperative Oncology Group (ECOG) performance status of =< 1 within 14 days prior to being registered for protocol therapy
* Females of childbearing potential and males must be willing to use an effective method of contraception (hormonal or barrier method of birth control; abstinence) from the time consent is signed until 4 weeks after treatment discontinuation
* Females of childbearing potential must have a negative pregnancy test within 7 days prior to being registered for protocol therapy

  * NOTE: Subjects are considered not of child bearing potential if they are surgically sterile (they have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are postmenopausal
* Females must not be breastfeeding
* Cohort A - T2, Transitional cell carcinoma (TCC) muscle invasive bladder cancer, (patients who are cisplatin ineligible, decline neoadjuvant and/or ineligible for neoadjuvant chemotherapy); must have histological proof of T2, muscle-invasive transitional cell carcinoma of the bladder with no evidence of metastatic; patient with any degree of fixation of the pelvic sidewall are not eligible
* Cohort B - Prostate cancer (Gleason 7 or less); must have histological proof of Gleason =< 7 with no evidence of metastatic disease (patient with any degree of extra-prostatic capsule extension are not eligible
* Cohort C - Renal cell carcinoma (> pT1b); must have radiologic suspicion or histological proof of clear cell renal cell carcinoma >= 4 cm with no evidence of metastatic disease; patient with any degree of tumor extension into the renal vein are not eligible; patients must be candidates for contrast-enhanced ultrasound (CEUS) imaging and agree to undergo this additional imaging technique
* Patients must be willing to undergo a biopsy of the cancerous tissue if one was not taken within the previous year, prior to drug initiation if tumor block is not available; biopsy must be done within 14 days of first planned drug dose
* Patients must be willing to undergo a radiologic scan (computed tomography [CT] or magnetic resonance imaging [MRI], depending on organ involved) after last drug dose and prior to minimally-invasive surgery
* Eligible for:

  * Cohort A: Robot-assisted radical cystectomy (RARC) as per the attending urologist
  * Cohort B: Robot-assisted radical Nephrectomy (RARN)/robot-assisted partial nephrectomy (RAPN) as per the attending urologist
  * Cohort C: RAPN as per the attending urologist
* No prior malignancy is allowed except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancers for which the patient has been disease-free for at least 5 years
* No treatment with any investigational agent within 30 days prior to being registered for protocol therapy
* No prior systemic chemotherapy for transitional cell carcinoma of the bladder (prior intravesical therapy is allowed); any other prior chemotherapy must have been completed > 5 years prior to initiation of therapy
* Prior radiation therapy is allowed provided that no radiation therapy was administered to the urinary bladder

  * NOTE: No radiation therapy within 28 days prior to being registered for protocol therapy; laboratory values must be obtained within 14 days prior to being registered for protocol therapy
* Total bilirubin < 2.0 X upper limit of normal (ULN)
* Aspartate aminotransferase (AST) =< 2.5 X ULN
* Alanine aminotransferase (ALT) =< 2.5 X ULN
* Serum Creatinine < 2.5 X ULN
* Absolute neutrophil count (ANC) > 1.5 X K/mm^3
* Platelets > 100 K/mm^3
* International normalized ratio (INR) =< 1.2
* There are currently no known concomitant medications that must be discontinued prior to administration of registration on study and for the duration of sEphB4-HSA
* No clinically significant infections as judged by the treating investigator
* No pleural or pericardial effusion of any grade
* No uncontrolled angina, congestive heart failure or myocardial infraction (MI) within 6 months prior to registration on study
* No diagnosed arrhythmias
* No abnormalities on pre-entry electrocardiogram, obtained within 28 days prior to being registered on study
* No history of diagnosed congenital bleeding disorders (e.g., von Willebrand's disease)
* No abnormalities no history of diagnosed acquired bleeding disorders within one year (e.g., acquired anti-factor VIII antibodies) of registration on protocol therapy
* No abnormalities no history of ongoing or recent (less than or equal to 3 months of registration on protocol therapy) significant gastrointestinal bleeding
* No ongoing anti-coagulation and/or anti-platelet therapies allowed
* Patients with diagnosed uncontrolled hypertension (> 150/90 mmHg) are to be excluded
* Patients with hypertension controlled with medications are allowed
* No evidence of gross hematuria
* No evidence of hydronephrosis
* No evidence of a history of a stroke or myocardial infarction within the last 6 months prior to study enrollment
* No evidence of a history of wound healing complications prior to study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-08-02 (Actual); Primary Completion 2020-01-28 (Actual); Study Completion 2021-11-15 (Actual)

PRIMARY OUTCOMES:
Feasibility, defined as the percentage of patients completing at least 3 doses of drug therapy without dose limiting toxicities (DLTs) and who are able to undergo minimally-invasive surgery as planned | Up to 30 days after the last dose of sEphB4-HSA
  Feasibility is defined for the purpose of this study as >= 90% of patients completing at least 3 doses of drug therapy without DLTs and are able to undergo minimally-invasive surgery as planned.
Incidence of adverse events graded according to CTCAE version 4 or the Clavien-Dindo classification | Up to 90 days post-surgery
  All observed adverse events and complications will be summarized in terms of type (organ affected or laboratory determination such as absolute neutrophil count), severity, and time of onset. Tables will be created to summarize these adverse events and complications, overall, by disease cohort, and by phase (neoadjuvant, during surgery, within 30 days post-operative, and days 31-90 post-operative).

SECONDARY OUTCOMES:
Complete pathologic response defined as no residual evidence of invasive disease at the time of cystectomy or nephrectomy | At the time of surgery
  Pathologic response rates will be calculated and 90% confidence intervals will be constructed.
Radiologic response as evaluated by Response Evaluation Criteria in Solid Tumors version 1.1 | Up to 30 days post-surgery
  Radiologic response rates will be calculated and 90% confidence intervals will be constructed.

CONTACTS AND LOCATIONS:
Overall Officials: David I Quinn, MD, Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States